CLINICAL TRIAL: NCT04773132
Title: Human Metabolic Flexibility: Its Role in Energy Regulation and Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, JeyaKumar Henry, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2014/01182
Record Dates: First submitted 2021-02-18; First posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Metabolic Flexibility
Keywords: BMR; P-ratio; Tissue partitioning
MeSH Terms: interventions — Diet, Protein-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low Protein Diet (Experimental): All subjects will be given a low protein/protein-free diet in order to deplete the label protein pool. The diet provided will meet the daily energy requirements of all the subjects.
  Interventions: Other: Low Protein

INTERVENTIONS:
Other: Low Protein — Low protein/protein-free diet for 3 days (Day 1, 2 and Day 3) in order to deplete the label protein pool. The diet provided will meet the daily energy requirements of all the subjects.

SUMMARY:
Obesity is commonly described as a consequence of excess calorie intake. Conventionally, the physiological variables that have been of extensive interest are food intake and energy expenditure. Despite decades of research on factors influencing intake and expenditure, to date, no compelling theory has been promulgated to explain why certain humans are more susceptible to weight gain than others. The investigators hypothesize that the measure of an individual's fraction of energy mobilized or deposited as protein (P-ratio), contributes towards an obese morphology and may essentially form a novel approach in understanding the etiology, management and treatment of obesity. In addition, there is a general perception that the consumption of sugar sweetened foods and beverages are one of the major causes of obesity. This study aims to understand metabolic flexibility and the glycemic index of diets in the etiology of obesity. Individual metabolic flexibility may be the key factor that predisposes an individual to obesity. This study is carried out to determine the P-ratio in human subjects.

DETAILED DESCRIPTION:
Obesity is commonly described as a consequence of excess calorie intake. Conventionally, the physiological variables that have been of extensive interest are food intake and energy expenditure. Despite decades of research on factors influencing intake and expenditure, to date, no compelling theory has been promulgated to explain why certain humans are more susceptible to weight gain than others. The investigators believe that a measure of an individual's metabolic flexibility towards an obese morphology is essential and forms a novel approach in understanding the etiology, management and treatment of obesity. Payne and Dugdale developed a simple model of energy balance, based on dividing the human body into four compartments, namely "fast" lean tissue (protein), "slow" lean tissue (protein), structural fat, and tissue fat. Notionally, these are considered to act as four separate compartments which interconnect with each other. Body weight is thus simply the sum of the four weights, and metabolic rate is the sum of the separate compartment rates. Any energy deficit in the "balancing compartment" is met by withdrawing tissues from the neighboring fat and lean (muscle) compartments in a proportion which is fixed for any individual. The observed human variability in both the susceptibility to gain weight or to lose weight efficiently on a calorie surplus or restricted diet is thus afforded by using the model developed by Payne and Dugdale for energy balance. P-ratio is calculated on the assumption that body protein is 16% nitrogen and has a metabolizable energy value of 16.7 kJ/g. Thus P-ratio can be calculated as: P- ratio= urinary nitrogen excretion x 6.25 x 16.7 / total energy expenditure. The regulatory control of energy-partitioning between protein and fat is highly variable between individuals, but constant within the same subject. It is this variability in tissue partitioning between lean (protein) and fat that is central to the regulation of body weight. This implies that for a given individual, there is a fixed partitioning of energy between lean (protein) and fat tissue when excess calories are consumed. Using the results of the classical study of human semi-starvation by Keys et al, Dugdale and Payne calculated the individual pattern of tissue mobilization (P-ratio) in these subjects. The P-ratio ranged from 0.03 to 0.60. On the basis of these data, they classified individuals into "metabolically lean" and "metabolically fat". A P-ratio of 0.03 means approximately 3% of the energy loss from this subject's body tissues was derived from protein catabolism and 97% from fat. Thus during excess calorie consumption, 3% of the calories will be deposited as protein and 97% as fat ("metabolically fat"). Similarly a subject with a P-ratio of 0.60 will deposit 60% calories as protein and only 40% as fat ("metabolically lean"). This stratification of "metabolic type" is a novel approach in obesity research, treatment and its management. The current method for the determination of P-ratio is based on subjects undergoing total starvation/fasting, e.g. complete food restriction, ad libitum water intake. This is a highly impractical approach. The investigator's proposal is to develop a more convenient and practical methodology to determine the P-ratio. An individual's Basal Metabolic Rate after a 10 hour overnight fast will approximate the denominator of the P-ratio. Henry et al reported a quantitative relationship between a fasting urine nitrogen loss (FUNL) and obligatory urinary nitrogen loss (OUNL), the ratio FUNL: OUNL remained close to 1.5. OUNL can be measured in urine when a subject is fed a protein free diet. With these two measures, the P-ratio of an individual can be estimated. OUNL is the protein lost in the urine when fed a zero or non-protein diet and fasting urinary loss is the nitrogen lost during starvation/ fasting (FUNL). The investigator's proposed study will be the first real-time study that will utilize the obligatory urine nitrogen loss and BMR to quantitate human P-ratio.

ELIGIBILITY:
Inclusion Criteria:

* Chinese Male or Female
* Age between 21-35 years
* Body mass index 17.5-32.0 kg/m2

Exclusion Criteria:

* People with major chronic disease such as heart disease, cancer or diabetes mellitus
* People with family history of diabetes
* People who have intolerances or allergies to study foods
* Individuals who are taking drugs known to affect glucose metabolism, body fat distribution, appetite, food intake or energy metabolism
* Individuals who are on a special diet or recently on a weight-lost diet
* Pregnant women

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2015-05-19 (Actual); Primary Completion 2016-04-01 (Actual); Study Completion 2017-12-11 (Actual)

PRIMARY OUTCOMES:
Weight | Day 1
  Kg
Waist Circumference | Day 1
  cm
Hip Circumference | Day 1
  cm
Body fat | Day 1
  Percentage
Estimated visceral adipose tissue area | Day 1
  cm2

SECONDARY OUTCOMES:
Height | Day 1
  cm

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No